CLINICAL TRIAL: NCT05331417
Title: Performance of a Bronchoscopic Score for Prediction of Tracheobronchial Herpes Simplex Virus Type 1 (HSV-1) Reactivation
Brief Title: Bronchoscopic Score for Prediction of Herpes Simplex-virus Type 1 (HSV-1) Reactivation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Other Study IDs: 06-AnIt-21
Record Dates: First submitted 2022-04-11; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Tracheobronchitis; Herpes Simplex Infection
Keywords: Bronchoscopy
MeSH Terms: conditions — Herpes Simplex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Patients with herpes-simplex infection requiring bronchoscopy — Due to the observational design of the study, no study-specific interventions are performed. The indication for bronchoscopy is determined by the responsible ICU physicians. Except for the above mentioned laboratory analyses, the treatment of the patients is completely guided by the responsible ICU physicians.
  Other Names: Observation

SUMMARY:
Tracheobronchial reactivation of HSV-1 is a common finding in critically ill patients and is associated with longer intensive care unit (ICU) stay and mechanical ventilation. At present it is unclear whether the presence of HSV-1 reactivation can be predicted by the clinical phenotype. In the present study, the performance of a bronchoscopic score of tracheobronchial inflammation for prediction of tracheobronchial HSV-1 reactivation is investigated

DETAILED DESCRIPTION:
Critically ill adult patients having a first diagnostic or therapeutic bronchoscopy are included. A standardized bronchoscopic score (values from 0 to 6) is assessed by an experienced ICU physician.

The score compounds are mucosal redness, mucosal swelling and vulnerability on contact. Compounds are quantified as "none" = 0, "some, disseminated" = 1, or "profound, ubiquitous" = 2 and added.

HSV-1 reactivation is detected by quantitative polymerase chain reaction (PCR) analysis of HSV-1-DNA from standardized bronchoalveolar lavage fluid.

In addition, HSV-1-DNA from blood and markers of immunocompetence (lymphocyte subtype count, monocyte count and Human Leukocyte Antigen - DR isotype (HLA-DR) expression, immunoglobulins) are measured for secondary analyses.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult patients (age ≥18 years) 2. Indication for bronchoscopy during intensive care unit stay 3. Written informed consent

Exclusion Criteria:

* 1. Solid organ transplantation 2. Present coronavirus disease 2019 (COVID-19) infection 3. Previous bronchoscopy during present hospital stay 4. Pregnancy 5. Known primary or secondary severe immunodeficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Bronchoscopic score for prediction of tracheobronchial HSV-1 reactivation | at study inclusion
  The score has values from 0 to 6, and for the primary analyses, HSV-1 reactivation is used as a binary variable (yes vs. no) dependent on the presence vs. absence of HSV-1-DNA in bronchoalveolar fluid.
  Sensitivity, specificity, positive and negative predictive values as well as best cut-off score values for prediction will be calculated

SECONDARY OUTCOMES:
Correlation of the bronchoscopic score value with quantitative tracheobronchial HSV-1-DNA load | day of study inclusion
Correlation of the bronchoscopic score value with quantitative blood HSV-1-DNA load | day of study inclusion
3. Correlation of tracheobronchial and blood HSV-1-DNA load with markers of immunosuppression (lymphocyte count, lymphocyte subgroups, monocyte count, monocyte HLA-DR expression, immunoglobulin concentration) | day of study inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Ertmer, MD, Study Chair — University Hospital Muenster, Dept. of Anesthesiology, Intensive Care Therapy and Pain Medicine
Locations (1):
- University Hospital Münster, Münster, Germany

IPD SHARING:
Plan to Share IPD: No